CLINICAL TRIAL: NCT00554073
Title: Whole Body Magnetic Resonance Angiography in Patients With Symptomatic Peripheral Ischemia: A Comparison Between 1.5 and 3T MRI-systems
Brief Title: Whole Body Magnetic Resonance Angiography in Ischemic Patients at 1.5 and 3T
Status: Suspended | Type: Observational
Why Stopped: It was not possible to perform 2 MRI studies in each patient due to practical problems. The study was not suspended due to safety issues.
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Yousef Nielsen, Department of Radiology, Copenhagen University Hospital Herlev
Other Study IDs: WB-angio herlev 2
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis; Intermittent Claudication; MRI
Keywords: Magnetic resonance; whole body; angiography; vasovist; gadofosveset; blood pool agent; 3T; 1.5T; Field strength
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the diagnostic performance of whole body magnetic resonance angiography (WB-MRA) using two different magnetic resonance scanners at a field strength of 1.5 and 3T. The hypothesis is that use of the 3T system gives superior signals from the investigated arteries, when compared with 1.5T.

DETAILED DESCRIPTION:
Atherosclerosis of the lower leg arteries is a common disease. Patients with this condition has symptoms of ischemia, for instance intermittent claudication (pain during exercise). Diagnosis of atherosclerosis in the legs is normally done with an interventional x-ray-based angiography (DSA- digital subtraction angiography). This is uncomfortable for the patient, and associated with risks of complications (bleeding, vascular damage, embolism).A novel approach to diagnosing atherosclerosis is the use of magnetic resonance angiography. A variant of this is the whole body magnetic resonance angiography(WB-MRA), that produce a picture of the arteries in almost the whole body (excluding the coronary arteries). WB-MRA has a number of advantages compared to DSA. It does not use ionizing radiation, is not invasive, uses a contrast medium with fewer side affects and finally gives a covers a great deal of the arteries in the body.

This study will compare WB-MRA with DSA in patients with symptoms of peripheral atherosclerosis in the lower legs.

All the patients will undergo arterial first pass whole-body MRA in the 3T-system. This will be followed by a WB-MRA steady state examination which can be performed because we use the intravascular contrast medium Vasovist, that has a prolonged intravascular life. The steady state examination will be performed in both the 3T and the 1.5T MR-system. Half the patients will have the steady state examination performed first in the 3T and then the 1.5T-system. The other half will go to the 1.5T-system first and then return to the 3T-system.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia (claudication, ischemic wounds) Referred to digital subtraction angiography (DSA)

Exclusion Criteria:

* Renal insufficiency (GFR < 30 ml/min)
* Contra-indications for MRI-examination (claustrophobia, metal-implants, pacemaker)
* Dementia
* Pregnancy/lactation
* Allergy to gadolinium based MRI contrast agents
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermittent claudication (pheripheral arterial disease)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2008-05; Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S Thomsen, Prof. MD., Study Chair — University Hospital at Herlev Copenhagen Denmark
Locations (1):
- Department of Radiology, Herlev University Hospital, Herlev Copenhagen, Herlev, Denmark